CLINICAL TRIAL: NCT00363077
Title: A Study to Evaluate the Immunogenicity, Safety and Reactogenicity of Adjuvanted Influenza Vaccine Candidate Compared to Fluarix™ (GlaxoSmithKline Biologicals) Administered Intramuscularly in Elderly Aged 60 Years and Older.
Brief Title: Study to Evaluate the Immunogenicity and the Safety of an Adjuvanted Influenza Vaccine Candidate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 107975
Record Dates: First submitted 2006-08-07; First posted 2006-08-15 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Influenza vaccine; Prophylaxis Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- GSK1247446A Group (Experimental): Subjects aged 60 years or older at the time of vaccination received 1 dose of the GSK1247446A vaccine adjuvanted with AS03. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK1247446A Group
- Fluarix Group (Active Comparator): Subjects aged 60 years or older at the time of vaccination received 1 dose of Fluarix™ vaccine. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix™

INTERVENTIONS:
Biological: GSK1247446A Group — Low dose influenza vaccine adjuvanted with AS03 compared
  Other Names: Low dose adjuvanted influenza vaccine
  Arms: GSK1247446A Group
Biological: Fluarix™ — GlaxoSmithKline (GSK) Biologicals' inactivated influenza split vaccine.
  Arms: Fluarix Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and the safety of the candidate vaccine compared to Fluarix™ administered intramuscularly in elderly aged 60 years and above

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and wil comply with the requirements of the protocol should be enrolled in the study.
* A male or female 60 years or older at the time of the first vaccination.
* Free of obvious health problems

Exclusion Criteria:

* Use of non-registered products
* Administration of immune-modifying drugs.
* Administration of vaccine 30 days before enrolment in study.
* Immunosuppressive or immunodeficient condition.
* Hypersensitivity to a previous dose of influenza vaccine
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality.
* History of confirmed influenza infection within the last 12 Months.
* Acute disease at the time of enrolment/vaccination.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-10-02; Primary Completion 2006-11-01 (Actual); Study Completion 2006-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 107975 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107975 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107975 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107975 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107975 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK1247446A Group | Fluarix Group
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1247446A Group | Fluarix Group | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (4.22) | 64.5 (4.18) | 64.4 (4.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 76
  Male | 37 | 37 | 74

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The 3 influenza strains assessed were A/New Caledonia, A/Wisconsin and B/Malaysia. The seropositivity cut-off assay was 1:10.
Time Frame: At Days 0 and 21
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects who received one dose of either study vaccine, for whom administration site of study vaccine was known, who did not receive a vaccine forbidden in the protocol and for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 74 | 74
titers
  A/New Caledonia, Day 0 | 45.3 [35.9 to 57.1] | 81.1 [61.5 to 106.8]
  A/New Caledonia, Day 21 | 116.4 [91.2 to 148.5] | 170.9 [132.7 to 220.3]
  A/Wisconsin, Day 0 | 28.8 [20.7 to 40.1] | 41.3 [29.1 to 58.6]
  A/Wisconsin, Day 21 | 251.9 [188.7 to 336.4] | 228.4 [168.5 to 309.6]
  B/Malaysia, Day 0 | 27.1 [21.8 to 33.6] | 31.6 [25.1 to 39.8]
  B/Malaysia, Day 21 | 161.6 [131.4 to 198.6] | 131.4 [105.8 to 163.1]

2. Primary Outcome: Number of Seroconverted Subjects Against 3 Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 3 influenza strains assessed were A/New Caledonia, A/Wisconsin and B/Malaysia.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 74 | 74
subjects
  A/New Caledonia | 21 | 12
  A/Wisconsin | 52 | 40
  B/Malaysia | 46 | 31

3. Primary Outcome: Number of Seroprotected Subjects Against 3 Strains of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:40. The 3 influenza strains assessed were A/New Caledonia, A/Wisconsin and B/Malaysia.
Time Frame: At Day 0 and Day 21
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 74 | 74
subjects
  A/New Caledonia, Day 0 | 40 | 54
  A/New Caledonia, Day 21 | 68 | 73
  A/Wisconsin, Day 0 | 35 | 44
  A/Wisconsin, Day 21 | 69 | 71
  B/Malaysia, Day 0 | 28 | 39
  B/Malaysia, Day 21 | 72 | 70

4. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease.
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 3 influenza strains assessed were A/New Caledonia, A/Wisconsin and B/Malaysia.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 74 | 74
fold increase
  A/New Caledonia | 2.6 [2.0 to 3.3] | 2.1 [1.6 to 2.8]
  A/Wisconsin | 8.7 [6.3 to 12.1] | 5.5 [4.0 to 7.6]
  B/Malaysia | 6.0 [4.6 to 7.8] | 4.2 [3.2 to 5.4]

5. Secondary Outcome: Geometric Mean of Influenza-specific Cluster of Differentiation (CD) 4 T-cells.
Description: The geometric mean was calculated for CD4 T-cells (per million CD4 T-cells) producing at least two different cytokines (All Doubles), at least CD40L, at least INF gamma (IFN-g), at least IL2 and at least TNF alpha (TNF-α).
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: cytokine-positive cells/million cells
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 73 | 73
cytokine-positive cells/million cells
  All Doubles, B/Malaysia, Day 0 [N=73;71] | 436.58 (348.81) | 451.35 (448.35)
  All Doubles, B/Malaysia, Day 21 [N=73;73] | 1555.92 (1060.11) | 736.15 (588.56)
  All Doubles, A/New Caledonia, Day 0 [N=73;71] | 322.57 (348.20) | 370.36 (408.19)
  All Doubles, A/New Caledonia, Day 21 [N=73;73] | 872.71 (662.32) | 510.86 (604.98)
  All Doubles, A/Wisconsin, Day 0 [N=73;71] | 37.33 (155.75) | 50.79 (212.97)
  All Doubles, A/Wisconsin, Day 21 [N=73;73] | 113.74 (412.68) | 72.43 (190.60)
  CD40L, B/Malaysia, Day 0 [N=73;71] | 424.07 (328.40) | 433.94 (406.20)
  CD40L, B/Malaysia, Day 21 [N=73;73] | 1409.79 (983.81) | 694.68 (550.36)
  CD40L, A/New Caledonia, Day 0 [N=73;71] | 317.25 (337.18) | 354.60 (399.44)
  CD40L, A/New Caledonia, Day 21 [N=73;73] | 786.97 (598.31) | 475.96 (576.45)
  CD40L, A/Wisconsin, Day 0 [N=73;71] | 36.53 (145.90) | 52.22 (208.27)
  CD40L, A/Wisconsin, Day 21 [N=73;73] | 97.23 (346.59) | 65.37 (168.16)
  IFN-g, B/Malaysia, Day 0 [N=73;71] | 265.46 (297.90) | 244.30 (377.07)
  IFN-g, B/Malaysia, Day 21 [N=73;73] | 1081.98 (840.54) | 530.64 (451.71)
  IFN-g, A/New Caledonia, Day 0 [N=73;71] | 225.76 (265.96) | 239.78 (285.26)
  IFN-g, A/New Caledonia, Day 21 [N=73;73] | 527.98 (522.30) | 407.10 (492.37)
  IFN-g, A/Wisconsin, Day 0 [N=73;71] | 24.45 (114.69) | 30.49 (83.91)
  IFN-g, A/Wisconsin, Day 21 [N=73;73] | 83.99 (365.27) | 38.46 (126.65)
  IL2, B/Malaysia, Day 0 [N=73;71] | 379.42 (318.77) | 382.48 (378.85)
  IL2, B/Malaysia, Day 21 [N=73;73] | 1297.82 (880.34) | 647.93 (508.83)
  IL2, A/New Caledonia, Day 0 [N=73;71] | 256.57 (307.83) | 220.62 (301.07)
  IL2, A/New Caledonia, Day 21 [N=73;73] | 652.75 (539.89) | 300.71 (502.30)
  IL2, A/Wisconsin, Day 0 [N=73;71] | 31.74 (130.05) | 53.93 (127.47)
  IL2, A/Wisconsin, Day 21 [N=73;73] | 89.97 (301.28) | 53.47 (148.09)
  TNF-α, B/Malaysia, Day 0 [N=73;71] | 332.83 (298.11) | 331.52 (383.96)
  TNF-α, B/Malaysia, Day 21 [N=73;73] | 1098.28 (869.02) | 532.81 (420.99)
  TNF-α, A/New Caledonia, Day 0 [N=73;71] | 219.03 (276.48) | 261.91 (369.60)
  TNF-α, A/New Caledonia, Day 21 [N=73;73] | 582.62 (506.95) | 317.96 (416.78)
  TNF-α, A/Wisconsin, Day 0 [N=73;71] | 23.29 (119.05) | 36.16 (190.06)
  TNF-α, A/Wisconsin, Day 21 [N=73;73] | 84.99 (308.52) | 44.97 (157.29)

6. Secondary Outcome: Geometric Mean of Influenza-specific Cluster of Differentiation (CD) 8 T-cells.
Description: The geometric mean was calculated for CD8 T-cells (per million CD8 T-cells) producing at least two different cytokines (All Doubles), at least CD40L, at least INF gamma (IFN-g), at least IL2 and at least TNF alpha (TNF-α).
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: cytokine-positive cells/million cells
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 73 | 73
cytokine-positive cells/million cells
  All doubles, B/Malaysia, Day 0 [N=72;69] | 7.91 (83.49) | 4.17 (70.59)
  All doubles, B/Malaysia, Day 21 [N=73;72] | 7.82 (95.80) | 3.74 (120.67)
  All doubles, A/New Caledonia, Day 0 [N=71;69] | 6.22 (233.32) | 7.31 (112.56)
  All doubles, A/New Caledonia, Day 21 [N=73;70] | 7.81 (191.24) | 4.40 (141.07)
  All doubles, A/Wisconsin, Day 0 [N=72;69] | 3.93 (82.82) | 6.79 (85.90)
  All doubles, A/Wisconsin, Day 21 [N=73;73] | 3.35 (56.70) | 2.79 (70.15)
  CD40L, B/Malaysia, Day 0 [N=72;69] | 2.20 (34.98) | 2.11 (36.15)
  CD40L, B/Malaysia, Day 21 [N=73;72] | 3.66 (45.91) | 1.98 (32.45)
  CD40L, A/New Caledonia, Day 0 [N=71;69] | 2.56 (113.11) | 5.34 (65.09)
  CD40L, A/New Caledonia, Day 21 [N=73;70] | 4.17 (93.16) | 2.11 (51.19)
  CD40L, A/Wisconsin, Day 0 [N=72;69] | 2.15 (53.59) | 2.70 (44.68)
  CD40L, A/Wisconsin, Day 21 [N=73;73] | 2.18 (39.28) | 2.11 (39.64)
  IFN-g, B/Malaysia, Day 0 [N=72;69] | 4.28 (56.03) | 2.71 (56.13)
  IFN-g, B/Malaysia, Day 21 [N=73;72] | 6.24 (74.51) | 3.53 (118.94)
  IFN-g, A/New Caledonia, Day 0 [N=71;69] | 5.67 (231.67) | 4.34 (97.73)
  IFN-g, A/New Caledonia, Day 21 [N=73;70] | 5.04 (174.85) | 3.98 (133.45)
  IFN-g, A/Wisconsin, Day 0 [N=72;69] | 2.84 (73.55) | 4.40 (69.48)
  IFN-g, A/Wisconsin, Day 21 [N=73;73] | 2.46 (44.69) | 1.98 (36.44)
  IL2, B/Malaysia, Day 0 [N=72;69] | 3.60 (92.44) | 2.12 (44.04)
  IL2, B/Malaysia, Day 21 [N=73;72] | 3.45 (60.32) | 2.44 (32.77)
  IL2, A/New Caledonia, Day 0 [N=71;69] | 2.48 (131.52) | 4.43 (60.02)
  IL2, A/New Caledonia, Day 21 [N=73;70] | 4.63 (125.59) | 2.44 (62.17)
  IL2, A/Wisconsin, Day 0 [N=72;69] | 1.93 (55.19) | 3.23 (61.15)
  IL2, A/Wisconsin, Day 21 [N=73;73] | 2.76 (45.28) | 2.55 (61.31)
  TNF-α, B/Malaysia, Day 0 [N=72;69] | 8.41 (83.63) | 4.29 (78.46)
  TNF-α, B/Malaysia, Day 21 [N=73;72] | 6.25 (91.95) | 3.90 (124.66)
  TNF-α, A/New Caledonia, Day 0 [N=71;69] | 6.07 (218.59) | 6.05 (114.14)
  TNF-α, A/New Caledonia, Day 21 [N=73;70] | 8.15 (171.91) | 5.50 (128.58)
  TNF-α, A/Wisconsin, Day 0 [N=72;69] | 3.12 (58.61) | 5.55 (92.14)
  TNF-α, A/Wisconsin, Day 21 [N=73;73] | 2.56 (49.21) | 2.33 (70.96)

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited Local Symptoms.
Description: Assessed solicited local symptoms were ecchymosis, pain, redness and swelling at injection site. Any = incidence of a particular symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling/ecchymosis = redness/swelling/ecchymosis spreading beyond 50 millimeters (mm) of the injection site. All solicited local symptoms were considered to be related to vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, on all subjects with the documented dose.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 75 | 75
subjects
  Any Ecchymosis | 1 | 1
  Ecchymosis > 50 mm | 1 | 0
  Any Pain | 57 | 25
  Grade 3 Pain | 1 | 0
  Any Redness | 14 | 8
  Redness > 50 mm | 4 | 0
  Any Swelling | 18 | 5
  Swelling > 50 mm | 3 | 1

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], headache, muscle aches and shivering. Any = incidence of a particular symptom regardless of grade intensity or relationship with the study vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0°C. Related = symptom considered by the investigator to have a causal relationship to study vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, on all subjects with the documented dose.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 75 | 75
subjects
  Any Arthralgia | 12 | 8
  Grade 3 Arthralgia | 0 | 0
  Related Arthralgia | 10 | 4
  Any Fatigue | 30 | 13
  Grade 3 Fatigue | 0 | 0
  Related Fatigue | 29 | 12
  Fever ≥ 37.5°C | 2 | 0
  Fever > 39.0°C | 0 | 0
  Related Fever | 2 | 0
  Any Headache | 28 | 10
  Grade 3 Headache | 0 | 0
  Related Headache | 24 | 7
  Any Muscle aches | 17 | 10
  Grade 3 Muscle aches | 1 | 0
  Related Muscle aches | 15 | 8
  Any Shivering | 10 | 3
  Grade 3 Shivering | 1 | 0
  Related Shivering | 9 | 3

9. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = any unsolicited AE regardless of intensity or relationship to vaccination. Grade 3 = unsolicited AE that prevented everyday activities. Related = unsolicited AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) post vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, on all subjects with the documented dose.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 75 | 75
subjects
  Subjects with any AE(s) | 31 | 22
  Subjects with grade 3 AE(s) | 1 | 0
  Subjects with related AE(s) | 11 | 7

10. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Related = SAE considered by the investigator to have a causal relationship to study vaccination.
Time Frame: During the entire study period (from Day 0 to Day 29)
Population: The analysis was performed on the Total Vaccinated cohort, on all subjects with the documented dose.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 75 | 75
subjects
  Subjects with any SAE(s) | 0 | 1
  Subjects with related SAE(s) | 0 | 0

ADVERSE EVENTS:
Time Frame: SAE(s): during the entire study (from Day 0 to Day 29); Solicited local and general symptoms: during the 7-day (Days 0-6) follow-up period after any vaccination; Unsolicited AE(s): during the 30-day (Days 0-29) follow-up period after any vaccination.
Arm/Group | GSK1247446A Group | Fluarix Group
Serious Adverse Events (participants affected / at risk) | 0/75 | 1/75
Other Adverse Events (participants affected / at risk) | 69/75 | 45/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1247446A Group (N=75) | Fluarix Group (N=75)
Coronary artery disease (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1247446A Group (N=75) | Fluarix Group (N=75)
Nasopharyngitis (Infections and infestations) | 7 | 4
Influenza like illness (General disorders) | 2 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pain (General disorders) | 57 | 25
Redness (General disorders) | 14 | 8
Swelling (General disorders) | 18 | 5
Arthralgia (General disorders) | 12 | 8
Fatigue (General disorders) | 30 | 13
Headache (General disorders) | 28 | 10
Muscle aches (General disorders) | 17 | 10
Shivering (General disorders) | 10 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.